CLINICAL TRIAL: NCT03706742
Title: STOP-HCC Evidence-Based Hepatocellular Cancer Prevention Through Treatment of Hepatitis C Virus Infection
Brief Title: STOP HCC: Mailed HCV Treatment Outreach Program for HCC Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Amit Singal, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: STU 072015-022
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis C; HepatoCellular Carcinoma
MeSH Terms: conditions — Hepatitis C; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients randomized to Group 1 will receive visit-based HCV screening, as offered by clinic providers as part of usual care. Providers must identify at-risk patients who are eligible for HCV screening, understand the benefits of screening in this population, and enter orders for HCV Ab testing. If the HCV antibody is abnormal, providers must order appropriate follow-up tests including HCV viral load to confirm HCV infection. Once HCV is confirmed, providers must refer the patients for fibrosis assessment and treatment evaluation. These efforts are augmented by an established best practice alert and health maintenance reminders.
- Mailed outreach (Active Comparator): Patients randomized to Group 2 will receive low literacy, written materials about HCV screening among baby-boomers in English and Spanish. The invitation will include patient-centered educational materials that discuss the risk of HCV in baby boomers and the benefits and risks of HCV screening. The invitation will include a phone number to schedule the HCV antibody blood test. Written materials will be developed and validated in Spanish using the Spanish Language Translation Resource. Once a potential subject is identified and randomized in Group 2, an outreach invitation will be mailed out. Shortly after the letter, a bilingual patient navigator will place a follow-up call to this potential subject. These follow-up calls will occur in the 2nd - 4th week after mailing invitations; up to three attempts in total will be made to reach the patient to facilitate HCC screening completion.
  Interventions: Behavioral: Mailed outreach

INTERVENTIONS:
Behavioral: Mailed outreach — The investigators will randomize all baby boomer patients (~12,000 patients) using a centrally maintained computer-generated list. Patients will be randomly assigned to one of two HCV screening strategies including: visit-based screening as part of usual care (Group 1) or mailed screening invitation outreach and centralized patient navigation (Group 2).
  Arms: Mailed outreach

SUMMARY:
Aim 1: The investigators will conduct a randomized controlled trial comparing two strategies to promote HCV screening, follow-up testing, and treatment among baby-boomers (i.e. persons born between 1945-1965): inreach with electronic medical record alerts and provider education vs. combination of inreach and provider education plus mailed outreach and patient navigation.

Aim 2: The investigators will evaluate patient navigation strategies to promote follow-up testing and treatment evaluation among non-baby boomer Parkland patients (i.e. born before 1945 or after 1965) who are either: a) HCV antibody positive but have not completed follow-up viral load testing or b) HCV viral load positive and who have not completed in-clinic treatment evaluation.

ELIGIBILITY:
Inclusion Criteria:

* born between 1945 and 1965
* ≥ 1 outpatient visit during 12 months prior to randomization at Parkland
* no prior HCV screening (prior HCV antibody, viral load, or genotype).
* any active medical coverage
* speaks Spanish or English

Exclusion Criteria:

* a life expectancy less than one year including end stage CHF, end stage COPD, metastatic cancer, and those who received a palliative care or hospice referral in the past year
* history of HCC.
* non-English or Spanish speakers
* no address or phone number on file

Ages: 53 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12386 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Hepatitis C Screening | 3 months
  Proportion with HCV Ab within 3 months of randomization

SECONDARY OUTCOMES:
Hepatitis C Screening | 12 months
  Proportion with HCV Ab within 12 months of randomization
Hepatitis C Confirmation | 3 months
  Proportion with HCV Viral Load within 3 months of positive antibody result
Hepatitis C Linkage to care | 6 months
  Proportion with clinic visit within 6 months of positive HCV Viral Load
Cost: Cost-per patient screened | 3 months
  The primary measure of costs will be the cost per Ab completion.
Cost: Cost per-HCV diagnosis | 12 months
  The primary measure of costs will be the cost per-patient diagnosed with HCV.

CONTACTS AND LOCATIONS:
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desai N, Rich NE, Jain MK, Blackwell JM, Murphy CC, Perryman P, McBryde J, Quirk L, Clark C, Villarreal D, Waljee AK, Gopal P, Singal AG. Randomized Clinical Trial of Inreach With or Without Mailed Outreach to Promote Hepatitis C Screening in a Difficult-to-Reach Patient Population. Am J Gastroenterol. 2021 May 1;116(5):976-983. doi: 10.14309/ajg.0000000000001085. PMID 33337657